CLINICAL TRIAL: NCT05350566
Title: Combined Effect of Exercise Intensity With Nutritional Supplementation on Skeletal Muscle Function
Acronym: NUTSPORT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne (Other)
Collaborators: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Principal Investigator, Nicolas Place, Principal Investigator, University of Lausanne
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2021-00373
Record Dates: First submitted 2022-04-14; First posted 2022-04-28 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Healthy Volunteers; Exercise Intensity; Neuromuscular Fatigue; Skeletal Muscle Adaptations
MeSH Terms: interventions — olive leaf extract

STUDY DESIGN:
Intervention Model Description: The design is a placebo-controlled, double blind, cross-over two-arm study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: One box containing the product and one containing the placebo will be labeled A or B. The code will be kept in a sealed envelope which will be revealed only at the end of the study or in case of an adverse event.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sprint interval training group (SIT group) (Experimental): The model of sprint interval training (SIT) consists of six 30 s all-out cycling bouts on a cycle ergometer, with 4 min rests between tests.
  Interventions: Dietary Supplement: Olive leaf extract; Dietary Supplement: Placebo
- Moderate intensity continuous training (MICT group) (Experimental): The moderate intensity continuous training (MICT) consists of 1h cycling on a cycle ergometer at 50% of the maximal aerobic power output
  Interventions: Dietary Supplement: Olive leaf extract; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Olive leaf extract — A capsule containing 250 mg of an olive leaf extract preparation will be swallowed with a glass of water before exercise.
Dietary Supplement: Placebo — A capsule containing 336 mg of cellulose microcrystalline will be swallowed with a glass of water before exercise.

SUMMARY:
The main objective of this study is to determine the effectiveness of a nutritional intervention (olive leaf extract) combined with a specific training session (MICT or SIT) on PDH activation (as well as other protein expressions) and exercise-induced muscle fatigue.

DETAILED DESCRIPTION:
Sprint interval training (SIT) is a form of interval training characterised by short bursts of intense exercise interspersed with rest periods. SIT is as, or more, effective than moderate intensity continuous training (MICT) for systemic and metabolic adaptations of muscles, despite a lower workload and shorter duration. However, the mechanisms underlying the metabolic response to SIT versus MICT are poorly understood. Our recent work (Zanou et al. 2021) suggests that increased pyruvate dehydrogenase (PDH) activity may explain why a SIT session led to greater changes in proteins involved in mitochondrial respiration compared to a MICT session.

Recently, it was found that a natural and commercially available compound based on olive leaf extract could stimulate resting mitochondrial bioenergetics by activating the mitochondrial calcium uniporter (MCU), which is involved in calcium transport across the mitochondrial membrane, directly controlling PDH activity. The main objective of this study is to determine the effectiveness of an acute nutritional intervention (olive leaf extract) combined with a specific training session (MICT or SIT) on PDH activation (as well as other protein expressions) and exercise-induced muscle fatigue.

Participants will be allocated to either a SIT (6 x 30 s all out sprints) or a MICT (1h at 50% maximal aerobic power) group and asked to come to the laboratory for five visits including one familiarization session with a triangular test for maximal aerobic power determination, the first experimental session during which they will realize the exercise with the product or a placebo and a session 24h after to assess skeletal muscle adaptations. Then after a 3 week wash-out period, they report to the laboratory for the fourth and fifth session, identical to the second and third sessions but with the other intervention (product or placebo). Muscle microbiopsies will be collected from the vastus lateralis muscle before, immediately after and 24 hours after exercise (MICT or SIT), while knee extensor neuromuscular function will be assessed at the same time points using voluntary and electrically-evoked contractions.

ELIGIBILITY:
Inclusion Criteria:

1. Being male (including females would necessitate increasing the number of included participants to consider sex as a variable which would burden the project too much).
2. Being aged between 18 and 40 years
3. Being healthy (The assessment will be done through a questionnaire and an interview/examination by a medical doctor if there is any doubts)
4. Being physically active, but not involved in any structured training program
5. Having stable dietary habits

Exclusion Criteria:

1. Having previous medical events that would put the participant at risk during the study
2. Ingesting caffeine on the experimental days
3. Not being currently treated for blood clotting problems
4. Taking aspirin or anti-coagulant drugs in the 48 hours preceding the experimental days in which muscle samples will be collected
5. Having allergy to xylocaine
6. Having food allergy

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2022-06-07 (Actual); Primary Completion 2022-12-07 (Actual); Study Completion 2022-12-07 (Actual)

PRIMARY OUTCOMES:
PDH dephosphorylation | before, immediately after and 24 hours after exercise completion
  protein involved in skeletal muscle metabolism
expression of OXPHOS proteins | before, immediately after and 24 hours after exercise completion
  proteins used as markers of oxidative phosphorylation complexes
expression of MCU protein | before, immediately after and 24 hours after exercise completion
  protein involved in the transport of Ca2+ in the mitochondria

SECONDARY OUTCOMES:
Maximal voluntary contraction force | before, immediately after and 24 hours after exercise completion
  Maximal force of the knee extensor muscles
Voluntary activation level | before, immediately after and 24 hours after exercise completion
  overall index of central fatigue induced by exercise
Peak doublet evoked at 100 Hz | before, immediately after and 24 hours after exercise completion
  overall index of peripheral fatigue induced by exercise
M-wave amplitude | before, immediately after and 24 hours after exercise completion
  index of neuromuscular excitability

CONTACTS AND LOCATIONS:
Locations (1):
- Bâtiment Synathlon, quartier UNIL-Centre, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Place N, Ivarsson N, Venckunas T, Neyroud D, Brazaitis M, Cheng AJ, Ochala J, Kamandulis S, Girard S, Volungevicius G, Pauzas H, Mekideche A, Kayser B, Martinez-Redondo V, Ruas JL, Bruton J, Truffert A, Lanner JT, Skurvydas A, Westerblad H. Ryanodine receptor fragmentation and sarcoplasmic reticulum Ca2+ leak after one session of high-intensity interval exercise. Proc Natl Acad Sci U S A. 2015 Dec 15;112(50):15492-7. doi: 10.1073/pnas.1507176112. Epub 2015 Nov 2. PMID 26575622
- [Background] Zanou N, Dridi H, Reiken S, Imamura de Lima T, Donnelly C, De Marchi U, Ferrini M, Vidal J, Sittenfeld L, Feige JN, Garcia-Roves PM, Lopez-Mejia IC, Marks AR, Auwerx J, Kayser B, Place N. Acute RyR1 Ca2+ leak enhances NADH-linked mitochondrial respiratory capacity. Nat Commun. 2021 Dec 10;12(1):7219. doi: 10.1038/s41467-021-27422-1. PMID 34893614